CLINICAL TRIAL: NCT02632877
Title: Efficacy of Pirfenidone Gel Combined With Modified Oxide Diallyl Disulfide (MODD) Versus Ketanserin for the Treatment of Diabetic Foot Ulcers
Brief Title: Efficacy of Pirfenidone Plus MODD in Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Cell Pharma (Other)
Responsible Party: Principal Investigator, Juan Armendáriz-Borunda, Head, Molecular Biology and Genomics Department, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBMMTG.14; ISSSTE/CEI/TR/2014/01 (Other: ISSSTE); Institute of Molecular Biology (Other: University of Guadalajara)
Record Dates: First submitted 2015-12-09; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: pirfenidone; Modified oxide diallyl disulfide (MODD); ketanserin; diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — pirfenidone; Ketanserin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pirfenidone with MODD (Experimental): Active ingredients: Pirfenidone 8% with modified oxide diallyl disulfide (MODD) 0.016%.
  Dosage form: gel. Dosage: standar finger tip unit (0.5g for an area of 100 to 120 square centimeters).
  Frequency and duration: topically applied every eight hours for 6 months.
  Interventions: Drug: Pirfenidone with MODD
- Ketanserin (Active Comparator): Active ingredients: Ketanserin 2%. Dosage form: gel. Dosage: standar finger tip unit (0.5g for an area of 100 to 120 square centimeters).
  Frequency and duration: topically applied every 12 hours for 6 months.
  Interventions: Drug: Ketanserin

INTERVENTIONS:
Drug: Pirfenidone with MODD — Patients with diabetic foot ulcer will be treated three times a day with a smooth layer (standar finger tip unit 0.5g for an area of 100 to 120 square centimeters) of KitosCell Q (Pirfenidone with MODD) in form of gel and the wound will be covered with a bandage.
  Other Names: KitosCell Q; 5-methyl-1-phenyl-2(1H)-pyridone with MODD
  Arms: Pirfenidone with MODD
Drug: Ketanserin — Patients will be administered ketanserin twice a day usign the standar finger tip unit (0.5g for an area of 100 to 120 square centimeters) and the wound will be covered with a bandage. This arm is a control for evolution of diabetic foot ulcer.
  Other Names: sufrexal
  Arms: Ketanserin

SUMMARY:
Diabetic foot ulcers (DFU) develop because of the interaction of predisposing factors like neuropathy, angiopathy and infection. Likewise, environmental factors like lesion hygiene, diet and life style.

DFU results as a complication in diabetic patients and it is the most common cause of non-traumatic foot amputation in people older than 50 years. Foot amputation decreases patients´ quality of life since only 33% of them will continue walking with the use of a prothesis.

However, 30% of patients subjected to amputation will die in the first year after surgery and by the 5th year, post-surgery 50% of them will need the amputation of the remaining body extremity.

According to the World Foundation for Diabetes, in Latin America there are 18 million people with Diabetes Mellitus Type 2 (DM2). This number will increase in the next 20 years to 30 million.

Medical expenses for diabetic patients are calculated to be around 8,000 million dollars, annually. In Mexico, according to the Mexican Federation for Diabetes there are 6.5-10 millions of diabetic patients.

Amputation due to DFU complications has many social and economic implications. In Mexico in 2011 diabetes mellitus complications were the principal cause of death in the institute of mexican social security (IMSS) population.

On the other hand, 5-methyl-1-phenyl-2-(1h)-pyridone (PFD) is considered an anti-inflammatory drug that promotes re-epithelization due to fibroblast stimulation, angiogenesis and vasculogenesis during tissue remodeling.

According to this, the investigators believe that PFD could play an important role in DFU resolution and for this reason, the investigators consider necessary to analyze the efficacy of 5-methyl-1-phenyl-2-(1h)-pyridone for the treatment of DFU since it has showed improvement in chronic skin ulcers in pilot studies.

Nowadays, DFU treatment includes management of metabolism, angiopathy and neuropathy along with broad-spectrum antibiotic therapy. However, several reports indicate it is insufficient for and adequate control of diabetic patients.

Then, it is important to develop efficient therapies for the treatment of DFU. In this context, Ketanserin (Sufrexal™) is a drug to induce scar formation. It has been demonstrated to decrease peripheral vascular resistance, platelet aggregation and improves hemorheologic parameters.

Topical administration of ketanserin has showed beneficial effects in inflammation, granulation and epithelization.

Since these two drugs have showed beneficial effects in tissue regeneration, the investigators believe it is important to compare their safety and efficacy for the treatment of DFU

DETAILED DESCRIPTION:
Subjects will be randomized using a random number table to distribute in the control (ketanserin) and the experimental group (PFD+MODD). Demographics data and medical history will be registered on a monthly basis, relative ulcer volume will be calculated by measuring the longest, widest and deepest ulcer side with sterile flexible graduated ruler. The ulcer will be classified according to Wagner scale and photographs will be taken. Ulcer area will be washed with aseptic solution (accua aseptic solution™) and a biopsy of around 10-15 mm3 will be taken from the middle of the ulcer using a scalpel blade. Patients in the experimental group will receive topical PFD+MODD (8% gel) three times a day and patients in control group will receive ketanserin (2% cream) twice a day. Both groups will apply the medicament for six months previous cleansing of the area. Biopsies will be taken at the beginning, at month one and month two. After this time, only photographs will be performed, and relative ulcer volume will be measured. 5 ml of blood will be taken at the beginning and the end of the study to measure general clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic for diabetic foot ulcer grade I to II according to Wagner scale
* Volunteer patients that accept to sign an informed consent letter
* Patients that agree to fill a clinical history, access to physical exploration and biochemical analysis samples, ulcer biopsy and photodocumentation of ulcer progress.
* Patients willing to sign a compliance letter to apply treatment as indicated by the principal investigator.

Exclusion Criteria:

* Patients with another chronic disease like venous insufficiency or cardiopathy.
* Patients with severe arteriopathy that do not have possibility to direct revascularization like the ones subject to graft tissue, plastics or stents positioning.
* Patients with severe arteriopathy that do not have possibility to indirect vascularization like the ones subject to sympathectomy .

Elimination criteria:

* Patients without adherence to treatment
* Patients that miss medical appointments
* Patients that show allergy to the 8% 5-methyl-1-phenyl-2-(1h pyridone gel and MODD or any of its components.
* Patients allergic to the 2% ketanserin gel or any of its components.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
assessing change of ulcerated area | 1, 2, 3, 4, 5, and 6 months
  mm3

SECONDARY OUTCOMES:
mRNA levels of collagen type I alpha (COL-1a) | 0, 1 and 2 months
  expression relative units
mRNA levels of Transforming growth factor 1-beta (TGFb-1) | 0, 1 and 2 months
  expression relative units
mRNA levels of Transforming growth factor 3-beta (TGFb-3) | 0, 1 and 2 months
  expression relative units
mRNA levels of Vascular endothelial growth factor (VEGF) | 0, 1 and 2 months
  expression relative units
mRNA levels of Tumor necrosis factor alpha (TNFa) | 0, 1 and 2 months
  expression relative units
mRNA levels of Hypoxia-inducible factor 1-alpha (HIF-1a) | 0, 1 and 2 months
  expression relative units
mRNA levels of Hypoxia-inducible factor 1-betha (HIF-1b) | 0, 1 and 2 months
  expression relative units
mRNA levels of Keratinocyte Growth Factor (KGF) | 0, 1 and 2 months
  expression relative units
mRNA levels of Matrix metalloproteinase-1 (MMP-1) | 0, 1 and 2 months
  expression relative units

CONTACTS AND LOCATIONS:
Overall Officials: Juan Armendariz-Borunda, PhD, FAASLD, Study Director — University of Guadalajara
Locations (2):
- Mexico (2):
  - Molecular Biology and Gene Therapy Institute, Guadalajara, Jalisco
  - Hospital Valentín Gómez Farías, Zapopan, Jalisco